CLINICAL TRIAL: NCT04633694
Title: Insect Protein - a New and Sustainable Protein Source to Maintain and Build Muscle
Brief Title: Insect Protein and Muscle Protein Signaling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: AP Moeller Foundation (Other); Beckett Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Proteinlab P4 Insect
Record Dates: First submitted 2020-08-10; First posted 2020-11-18 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Sarcopenia
Keywords: mTORC metabolomics,; Western blotting; Real time quantitative polymerase chain reaction; Nuclear magnetic resonance; Liquid chromatography-mass spectrometry
MeSH Terms: conditions — Sarcopenia | interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: A parallel 3 armed study, each arm with a different protein type
Who Masked: Participant, Care Provider
Masking Description: The project leader are responsible for the masking while all other persons involved in the project do not know the protein source given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Insect protein (Experimental): The participants are are given insect protein
  Interventions: Dietary Supplement: insect, pea or whey protein
- Pea protein (Experimental): The participants are are given pea protein
  Interventions: Dietary Supplement: insect, pea or whey protein
- Whey protein (Experimental): The participants are are given whey protein
  Interventions: Dietary Supplement: insect, pea or whey protein

INTERVENTIONS:
Dietary Supplement: insect, pea or whey protein — The protein powder is dissolved in 400 mL water and given relative to lean body mass, 0.25 g protein pr kg lean body mass.

SUMMARY:
Randomized parallel study investing the effect of intake of different protein sources (whey, insect and pea) on the muscle protein synthesis. Activation of the signaling pathway leading to muscle protein synthesis is investigated by western blotting and Real time quantitative polymerase chain reaction (qPCR or PCR). Urine, blood and muscle is moreover investigated by metabolomics analysis.

DETAILED DESCRIPTION:
Background:

Sarcopenia is a syndrome highly prevalent in the older population, characterized by muscle loss and a decrease in muscle strength. This leads to loss of physical function, decreased life quality and well-being and an increased risk of early death. Research has shown that both ingestion of protein and physical activity is able to diminish the loss of muscle mass during aging and thereby reduce the prevalence of sarcopenia and diminish the consequence of the disease. This study will investigate if more sustainable protein sources of good quality can increase the muscle protein synthesis and thereby prevent sarcopenia.

Aim:

The aim of this project is to investigate the effects of insect protein on the stimulation of muscle protein synthesis. The effects of protein will both be studied alone and in combination with exercise in perspective of preventing loss of both muscle mass and muscle strength. The potential of insect protein will be elucidated by comparison with other alternative plant-based protein sources in this case pea protein. In addition, whey protein will be included as a positive control as it may be regarded as the most established dietary protein source combatting muscle loss.

Method:

Young(18-30 years old) healthy men (n=60) are randomized in 3 groups to ingest either insect protein, pea protein or whey protein. Urine are collected 24 hours prior to the experiment while a blood sample and a muscle biopsy is collected at the beginning of the study. The subjects are instructed to perform one-leg exercise (knee extension, 5 sets of 10 repetitions, 10 repetitions-maximum) after which the subjects ingest the assigned protein bolus. Urine and blood samples are collected in the following hours and one muscle biopsy is collected from both the exercised and the non-exercised leg at 3 hours after protein ingestion. The expression of messenger RNA (mRNA) and protein related to the mTORC pathway in the muscle is investigated by qPCR and western blotting. In addition, metabolites in urine, blood plasma and muscle tissue are investigated by metabolomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18-30 year
* able to read and understand danish

Exclusion Criteria:

* smoking
* resistance training more than 1 time pr month
* endurance training more than 2 hours pr week
* Allergy toward shellfish, house dust mites or the protein sources.
* knee problems effecting the exercise
* weight change more than 5 kg the last half year
* medicine which can effect the protein turnover
* Disease in joint, or muscle as well as metabolic diseases.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Expression and phosphorylation of signaling proteins and their mRNA by Western Blotting and PCR | 4 hours
  Change in expression and phosphorylation of signaling proteins and the mRNA related the muscle protein synthesis.
Blod and urine metabolism by NMR | 4 hours
  Both blod and urine are analysed by nuclear magnetic resonance (NMR) metabolomics to enlighten changes in the metabolites.
Muscle metabolism by NMR | 3 hours
  The muscle metabolites are quantified before intervention, after protein and after protein end exercise.

SECONDARY OUTCOMES:
BMI | 1 hour
  Control parameter between groups. Measured before the study day.
General physical activity | 3 months
  in the last 3 month. Self-reported through a questionnaire.
Blood glucose | 4 hours
  Blood glucose measured at 7 time points over the 4 hour period.
Blood Insulin | 4 hours
  Blood insulin is measured at 7 time points over the 4 hour period.
Food intake, calories and distribution of macro nutrients. | 1 day
  Control parameter between groups. Self-reported diet report.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health,, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
All analysis will be performed within the research team.

REFERENCES:
- [Derived] Lanng SK, Oxfeldt M, Pedersen SS, Johansen FT, Risikesan J, Lejel T, Bertram HC, Hansen M. Influence of protein source (cricket, pea, whey) on amino acid bioavailability and activation of the mTORC1 signaling pathway after resistance exercise in healthy young males. Eur J Nutr. 2023 Apr;62(3):1295-1308. doi: 10.1007/s00394-022-03071-y. Epub 2022 Dec 19. PMID 36536114